CLINICAL TRIAL: NCT04701801
Title: Correlation of Preoperative Anxiety With Early Postoperative Cognitive Dysfunction in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gizem Fariz, research assistant, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2020-10/850; 2020-10/850 (Other: Ankara Oncology hospital clinical research ethics committee)
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Cognitive Dysfunction; Preoperative Anxiety
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MoCA test — Preoperative MoCA test and State-Trait Anxiety Inventory Test (STAI FORM ) questionnaire form will be filled in female patients between the ages of 18-65 by making a one-on-one interview with the patient and the MoCA test will be applied in the early postoperative period (1st week) to ensure its relationship with POCD will be checked.

SUMMARY:
Breast cancer is the most common type of cancer in women. Anxiety and depression often accompany the treatment phase of oncology patients.

Since both anxiety and depression are associated with increased inflammatory activity, these preoperative symptoms may predispose patients to the development of postoperative neurocognitive dysfunction.

The aim of this study is to reveal the correlation of preoperative anxiety with early postoperative cognitive dysfunction in patients with breast cancer who will undergo surgery.

DETAILED DESCRIPTION:
During the treatment of oncological disease, %13-19 of these patients show symptoms of anxiety and depression.Although many factors affect the development of postoperative cognitive dysfunction, there are several well-known risk factors and are thought to be due to increased inflammatory activity. Inflammation and immune dysfunction are common in oncological patients. It has also been reported that the presence of increased central nervous system inflammatory reactivity affects cognitive function.Since both anxiety and depression are associated with increased inflammatory activity, these preoperative symptoms may predispose patients to the development of postoperative neurocognitive dysfunction.

Postoperative cognitive dysfunction is an unwanted postoperative condition and is thought to be particularly relevant to elderly patients. Most studies in the literature have focused on the elderly. However, younger patients tend to experience more anxiety and depression during cancer treatment.

Studies indicate that age is inversely correlated with emotional distress and younger patients tend to experience higher levels of anxiety during diagnosis and treatment.

Also, younger patients have more limited life experiences to help them cope with such traumatic situations. The preoperative anxiety rate was found twice as high in female patients compared to male patients. Younger patients with bone cancer, breast cancer, and prostate cancer were three times more likely to report anxiety among the tumor groups than older patients.

Although the definition, degree and duration of postoperative cognitive dysfunction have been well researched, the effect of preoperative anxiety on the development of postoperative cognitive dysfunction has not been studied in detail.

Patients who are scheduled for elective breast surgery will be included in the study, who are informed and agree to participate in the study.

From the beginning of the study, consecutive patients will be included in the study.Preoperative MoCA test and State-Trait Anxiety Inventory Test (STAI FORM) questionnaire form will be filled in with the patient through one-on-one interview and in the early postoperative period. After the test ASA scores, age, comorbidities, demographic data, education levels, duration of anesthesia and surgery, and vital parameters will be recorded.

(1st week) MoCA test will be applied and its relationship with POCD will be checked.

Patients with preoperative MoCA score (M0) 21/30 points and above; It will be re-evaluated on the 7th postoperative day (M1) and a 4 unit decrease in M1 score from M0 score will be considered as POCD.

The correlation between preoperative anxiety level and early postoperative cognitive dysfunction (POCD) will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Should be female
2. Should be between 18-65 years old
3. Diagnosed with breast cancer
4. Scoring 21 or above in the MoCA test,
5. Patients under general anesthesia
6. Are decided to have Total Mastectomy, Modified Radical Mastectomy or Breast Conserving surgery
7. Having a risk score of The American society of Anesthesiologists (ASA) risk score 3 and below

Exclusion Criteria:

1. Cerebral ischemia or hemorrhage history
2. Clinical diagnosis of Neurodegenerative disease
3. Clinical diagnosis of carotid stenosis,
4. The score 20 or less in the Moca test,
5. Carotid endarterectomy history
6. Aneurysm surgery history
7. Alcohol addiction
8. Clinical diagnosis of psychiatric disease
9. Cervical surgery history
10. Inability to comply with the questionnaire or study
11. Chemotherapy history

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The preoperative anxiety rate was found twice as high in female patients compared to male patients.
Study Population: Female patients aged 18-65 years who are scheduled for elective surgery due to breast malignancy who meet the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Determining the preoperative anxiety level and evaluating the difference between the preoperative moca test and the moca test performed on the postoperative 7th day (early period) | 7th postoperative day
  The researcher will perform the neurocognitive level with a face-to-face interview with the moca test before surgery. In the postoperative period, the test will be repeated on the 7th day.
  If the moca test is above 21, it will be considered normal. and the patient will be enrolled.
  A decrease of 4 units in the moca test on the 7th postoperative day will be considered as postoperative cognitive dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr.Abdurrahman Yurtaslan Ankara Oncology Education and Research Hospital clinic of Anesthesiology and Reanimation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Linden W, Vodermaier A, Mackenzie R, Greig D. Anxiety and depression after cancer diagnosis: prevalence rates by cancer type, gender, and age. J Affect Disord. 2012 Dec 10;141(2-3):343-51. doi: 10.1016/j.jad.2012.03.025. Epub 2012 Jun 21. PMID 22727334
- [Background] Alam A, Hana Z, Jin Z, Suen KC, Ma D. Surgery, neuroinflammation and cognitive impairment. EBioMedicine. 2018 Nov;37:547-556. doi: 10.1016/j.ebiom.2018.10.021. Epub 2018 Oct 19. PMID 30348620
- [Background] Peng L, Xu L, Ouyang W. Role of peripheral inflammatory markers in postoperative cognitive dysfunction (POCD): a meta-analysis. PLoS One. 2013 Nov 13;8(11):e79624. doi: 10.1371/journal.pone.0079624. eCollection 2013. PMID 24236147
- [Background] Camacho A. Is anxious-depression an inflammatory state? Med Hypotheses. 2013 Oct;81(4):577-81. doi: 10.1016/j.mehy.2013.07.006. Epub 2013 Jul 26. PMID 23891039
- [Background] Carlson LE, Angen M, Cullum J, Goodey E, Koopmans J, Lamont L, MacRae JH, Martin M, Pelletier G, Robinson J, Simpson JS, Speca M, Tillotson L, Bultz BD. High levels of untreated distress and fatigue in cancer patients. Br J Cancer. 2004 Jun 14;90(12):2297-304. doi: 10.1038/sj.bjc.6601887. PMID 15162149